CLINICAL TRIAL: NCT03315728
Title: Transformation of Indigenous Primary Healthcare Delivery: Enhancement and Adaptation of Community-driven Innovations and Scale-up Toolkits
Brief Title: Pathways for Health Equity Quality Improvement Strategy
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AstraZeneca (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Stewart Harris, Principal Investigator, Western University, Canada
Other Study IDs: R2722A59
Record Dates: First submitted 2017-10-03; First posted 2017-10-20 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus Type 2 With Hyperglycemia
Keywords: Quality improvement; Indigenous; First Nation; Participatory; Diabetes; Chronic Disease
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality Improvement Strategy: First Nations communities partners are a diverse group of Indigenous communities reflecting wide variation in contextual factors: healthcare delivery and funding models; population size; remoteness; governance structures; and access to primary, secondary and tertiary care. Four diverse communities will partner in the program (two in Ontario and two in Atlantic Canada). All four communities will undertake an 18- month Quality Improvement Strategy intervention where they develop community-driven and culturally-relevant initiatives to improve diabetes care and management in their community
  Interventions: Other: Quality Improvement Strategy

INTERVENTIONS:
Other: Quality Improvement Strategy — Quality improvement strategy The 18 month Quality Improvement Strategy includes 3 months preparation, 12 months intervention, 3 months local knowledge translation. The intervention includes Readiness Consultations to assist in understanding available resources to address and adopt diabetes and chronic disease prevention and care strategies. Community teams receive a series of 3 workshops (in-person/virtual) followed by action periods where the team carry out and evaluate PDSAs they develop to improve diabetes care. Coaching is provided by Western during the 3-4 month action periods. FNDSS is a webbased secure community portal system for communities to develop a diabetes registry/surveillance system and generate reports and plan QI initiatives.

SUMMARY:
The PATHWAYS for Health Equity research program builds on the 5-year FORGE AHEAD Indigenous diabetes quality improvement research program (2013 - 2017).

PATHWAYS for Health Equity, a 3-year research program (2017 - 2019), is a great opportunity to continue our important collaborative diabetes quality improvement research with an increasing number of Indigenous partnering communities and researchers and key stakeholders (collaborators, policymakers and knowledge-users). Four partnering First Nations communities will join the Pathways program to develop community-driven quality improvement initiatives championed by a Community Facilitator and supported by a Community Data Coordinator.

DETAILED DESCRIPTION:
GOAL

To improve the health and health equity of Indigenous peoples by strengthening the effectiveness, sustainability and scalability of a promising community-driven and culturally-relevant quality improvement strategy through meaningful conversations and engagement with our community partners.

OBJECTIVES

1. Engage community partners and key stakeholders to support meaningful participation and leadership
2. Review, improve and adapt the diabetes quality improvement strategy with community partners
3. Evaluate the effectiveness of the adapted diabetes quality improvement strategy
4. Develop community-driven plans for sustainability and scale-up for the adapted diabetes quality improvement strategy

WHY IS PATHWAYS IMPORTANT?

In Canada, there are significant inequalities between the health status of Indigenous peoples and the general population concerning diabetes. Community-driven initiatives using promising diabetes quality improvement strategies can potentially reform local healthcare in Indigenous communities and improve care for those living with diabetes.

WHAT IS INVOLVED IN PATHWAYS?

Community-based champions called Community Facilitators and Community Data Coordinators will be trained to provide leadership and support to community-based teams to make priority improvements to diabetes programs/ services and clinical care. The 18-month quality improvement intervention includes:

* educational workshops on diabetes and quality improvement
* support, communication, and coaching for action planning and quality improvement
* readiness consultation tools
* diabetes registry & surveillance system

An evaluation consisting of interviews and questionnaires may be used to understand the process of adapting the diabetes quality improvement strategy to each community's context and factors that influence the program's success.

Our strong, multidisciplinary and cross-jurisdictional PATHWAYS Team includes Indigenous community representatives and healthcare providers, nonIndigenous healthcare providers, clinician scientists and academic researchers, as well as policy decision-makers and knowledge-user organizations.

The timely program will provide community leaders and knowledge-users with policy recommendations and a quality improvement strategy that can be implemented, sustained and spread to Indigenous community settings and regions across Canada and internationally.

COMMUNITY PARTNERS

Four community partners will be engaged and will partner in the Pathways program (two in Ontario and two in Atlantic Canada). Formal Community Research Agreements will represent participation and partnership.

ELIGIBILITY:
Inclusion Criteria:

Indigenous Communities in Canada:

1. On-reserve community
2. Community Band Council approval to participate and collaboration
3. Community healthcare facility approval or willingness to participate including both prevention and management/treatment arms if separate
4. Signed Community Research Agreement (including Financial Agreement) by the custodian of community medical charts, health leadership, and community leadership (if required). Access to community medical charts is required for FNDSS

Patient Chart Inclusion Criteria for chart audit component:

1. Age 18 or older.
2. Diagnosed with type 2 diabetes

Exclusion Criteria:

Indigenous Communities:

1. Communities that are unlikely to comply with the protocol (uncooperative attitude, unlikelihood of completing the program)
2. Healthcare facility unwilling to participate or uncooperative.

Patient Chart Exclusion Criteria for chart audit component:

1. Less than 18 years old
2. Diagnosed with type 1 or gestational diabetes
3. Life expectancy is less than 6 months
4. Inactive patient (no clinic visit in the last 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First Nation Community Partners, their local leadership, members (inclusive of Elders, youth, and women), and those who provide healthcare and prevention programs to community members, will be involved on the Implementation Research Team and lead enhancements/ adaptations of the QI Strategy prior to implementation, AND oversee the intervention and research in each of the communities. Community partners are a diverse group of Indigenous communities reflecting a wide variation in contextual factors including healthcare delivery and funding models, population size, remoteness, governance structures, access to primary, secondary and tertiary care, and readiness to participate in a QI program.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Understand the influence of community context on the implementation of the QI Strategy as assessed by the Consolidated Framework for Implementation Research | November 2017 - April 2019
  Qualitative information will be collected by interviews or focus groups to understand how context influences the implementation of the QI strategy. Questions on the interview are guided by the Consolidated Framework for Implementation Research, which includes questions on intervention characteristics, outer community setting, inner community setting, characteristics of individuals/teams, and implementation processes.

SECONDARY OUTCOMES:
Glycated hemoglobin (A1C) | November 2017 - April 2019
  Improvement in A1C will be assessed using the community's FNDSS portal.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Harris, MD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no sharing of individual participant data.

REFERENCES:
- See also: Description of Pathways for Health Equity Website — https://www.uwo.ca/diabetesalliance/indigenous/soar/index.html